CLINICAL TRIAL: NCT04088448
Title: The Antidiabetic Metformin as a Novel Adjunct to Antidepressants in Major Depressive Disorder Patients: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Antidiabetic Metformin as a Novel Adjunct to Antidepressants in Major Depressive Disorder Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0056/2018
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Fluoxetine 20 mg capsule once daily for 12 week plus placebo tablet once daily for 12 weeks
  Interventions: Drug: Placebo oral tablet
- Metformin group (Experimental): Fluoxetine 20 mg capsule once daily for 12 week plus Metformin 1000 mg XR tablet once daily for 12 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Placebo oral tablet — Fluoxetine 20 mg capsule plus Placebo tablet administered once daily after food
  Arms: Control group
Drug: Metformin — Fluoxetine 20 mg capsule plus Metformin 1000 mg extended release tablet administered once daily after food
  Arms: Metformin group

SUMMARY:
The aim of our study was to test whether the combined administration of the SSRI fluoxetine and metformin, a drug improving metabolic profile and therefore potentially able to mimic the influence of supportive living conditions on treatment outcome, results in an improved antidepressant efficacy compared with fluoxetine alone.

DETAILED DESCRIPTION:
Selective Serotonin Reuptake Inhibitors (SSRIs) represent the standard treatment for Major Depressive Disorder (MDD). However, their efficacy is variable and incomplete. In order to explain, at least in part, such variable efficacy, we have shown that SSRI administration does not affect mood per se but, by enhancing neural plasticity, amplifies the influence of the living conditions on mood. Consequently, in a favorable environment, SSRI treatment leads to a reduction of symptoms while, in stressful conditions, it could lead to a worse prognosis. Here, we test the hypothesis that, given the clear association between living conditions and metabolic profile, the modulation of the latter may mimic the effect of the environment on SSRI outcome, determining treatment efficacy.

Metformin is widely used as a first line treatment for patients with type 2 diabetes mellitus for more than 60 years for the reduction of hepatic glucose output and increase of the insulin mediated utilization of glucose. Previous studies demonstrated that metformin can rapidly cross the blood brain barrier and has several beneficial effects in the brain such as anti-inflammatory and neuroprotective effects. Furthermore, metformin, along with its anti-glycemic effects, has been documented to possess anti-depression effects in patients with type 2 diabetes. In Guo's study, 58 participants diagnosed with depression and type 2 diabetes were divided into two groups: one treated with metformin and the other with a placebo for 24 weeks. Analysis of MADRS and HRSD-17 scores showed that metformin significantly reduced MADRS scores and HRSD-17 scores. Metformin administration improves depressive symptoms in type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Eighty adult outpatients with the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of MDD based on a MINI Neuropsychiatric Interview (MINI) (American Psychiatric Association., 2000; Sheehan et al., 1998), without psychotic features and a total 17 item HAM-D score of at least 18 with item 1 (depressed mood) scored 2 or greater were eligible (Hamilton, 1960).
* Patients were requested to be free of all the psychotropic and anti-inflammatory medications for at least 4 weeks before participating in the study.

Exclusion Criteria:

* Patients with bipolar I or bipolar II disorder
* Patients with personality disorders
* Patients with eating disorders
* Patients with substance dependence or abuse
* Patients with concurrent active medical condition
* Patients with history of seizures
* Patients with history of receiving Electroconvulsive therapy (ECT)
* Patients with diabetes and other inflammatory disorders
* Patients with allergy or contraindications to the used medications
* Patients with finally pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Effect on Hamilton Depression rating scale score (HAM-D score) | Baseline to week 12
  The principal measure of the outcome was the 17-items HAM-D. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-13 suggest mild depression, 14-17 moderate depression and scores over 17 are indicative of severe depression. Remission is defined as HAM-D total score ≤ 7 (primary outcome). Treatment response is defined as ≥ 50% drop in the HAM-D total score.

SECONDARY OUTCOMES:
TNF-α | Baseline to week 12
  Serum level of tumor necrosis factor alpha (TNF-α)
BDNF | Baseline to week 12
  Serum level of brain derived neurotrophic factor (BDNF),
CRP | Baseline to week 12
  Serum level of C-Reactive Protein
IGF-1 | Baseline to week 12
  Serum level of Insulin-Like Growth Factor

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
URL: https://link.springer.com/article/10.1007/s13311-020-00878-7

REFERENCES:
- [Derived] Abdallah MS, Mosalam EM, Zidan AA, Elattar KS, Zaki SA, Ramadan AN, Ebeid AM. The Antidiabetic Metformin as an Adjunct to Antidepressants in Patients with Major Depressive Disorder: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial. Neurotherapeutics. 2020 Oct;17(4):1897-1906. doi: 10.1007/s13311-020-00878-7. PMID 32500486 (Retraction: PMID 36071262 Neurotherapeutics. 2022 Sep;19(5):1687)
- See also: The Antidiabetic Metformin as an Adjunct to Antidepressants in Patients with Major Depressive Disorder: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial — https://link.springer.com/article/10.1007/s13311-020-00878-7